CLINICAL TRIAL: NCT05894837
Title: Serplulimab in Combination With Regorafenib and Hepatic Artery Bicarbonate Infusion for Third-line Treatment in Patients With Colorectal Cancer and Liver Metastases: a Single-center, Single-arm, Phase 2 Trial
Brief Title: Serplulimab+Regorafenib +Hepatic Artery Bicarbonate Infusion in Patients With Colorectal Cancer and Liver Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-034
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Colorectal Cancer; Regorafenib; hepatic artery bicarbonate infusion; Serplulimab
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab in combination with Regorafenib and hepatic artery bicarbonate infusion (Experimental): Serplulimab: once every two weeks; Regorafenib: from the first day to the 21th day; hepatic artery bicarbonate infusion: once every four weeks
  Interventions: Drug: Serplulimab+Regorafenib; Drug: Hepatic Artery Bicarbonate Infusion

INTERVENTIONS:
Drug: Serplulimab+Regorafenib — Serplulimab: once every two weeks; Regorafenib: from the first day to the 21st day
Drug: Hepatic Artery Bicarbonate Infusion — hepatic artery bicarbonate infusion: once every four weeks

SUMMARY:
A single-center, single-arm, phase 2 trial of Serplulimab in combination with Regorafenib and hepatic artery bicarbonate infusion for third-line treatment in patients with colorectal cancer and liver metastases. A total of 30 patients are planned to be enrolled.

DETAILED DESCRIPTION:
This is a single-center, single-arm, phase 2 trial. Enroll 30 patients with colorectal cancer and liver metastases and failure of standard therapy. Administer serplulimab intravenously(once every two weeks)in combination with regorafenib(from the first day to the 21th day) and hepatic artery bicarbonate infusion (once every four weeks). Medication must be discontinued until disease progression, intolerable toxicity, informed consent is withdrawn, or investigator judgment is made. The primary endpoint is objective response rate (ORR), and secondary endpoints are progression-free survival (PFS), overall survival (OS), and adverse effects (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above, male or female;
2. Patients with colorectal cancer and liver metastases who strictly conform to the clinical diagnostic criteria of "Chinese Guidelines for Diagnosis and Treatment of Colorectal Cancer (2020 Edition)" or who have been confirmed by histopathology or cytology;
3. At least 1 measurable intrahepatic lesion;
4. Child-Pugh liver function rating: A or good B (≤7 points) ;
5. No local treatment including radiotherapy, surgical excision and ablation was performed before interventional therapy;
6. No other malignant tumors;
7. ECOG score within one week before enrollment: 0-1;
8. Predicted survival ≥24 weeks;
9. The major organs are functioning normally; the following criteria are met: Blood examination: a) HB≥90 g/L；b) ANC≥1.5×109/L；c) PLT≥80×109/L; Biochemical examination: a) ALB ≥29 g/L；b) ALT and AST<5ULN；c) TBIL ≤1.5ULN；d) Creatinine≤1.5ULN；(Only one of the two measures of albumin and bilirubin in the Child-Pugh rating can be a score of 2); Thyroid function tests are within normal range；
10. Women of childbearing age must already be using reliable contraception or have had a pregnancy test (serum or urine) with negative results within 7 days prior to inclusion and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last test drug administration；
11. The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up；

Exclusion Criteria:

1. There is a contraindication of anti-PD-1 monoclonal antibody therapy;
2. With other uncured malignancies, except for cured basal cell carcinoma of the skin and cervical carcinoma in situ;
3. Patients who are preparing for an organ transplant or have had an organ transplant in the past；
4. Ascites with clinical symptoms that require therapeutic abdominal puncture or drainage, or Child-Pugh score > 2；
5. Patients with high blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg) who cannot be reduced to the normal range by antihypertensive medication；
6. Patients with grade Ⅱ or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450 ms for males and 470 ms for females); A history of symptomatic ischemic or hemorrhagic cerebrovascular disease；
7. Having multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction, which significantly affects drug administration and absorption)；
8. Patients with a history of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within the past 6 months, such as esophageal varicose veins with bleeding risk, locally active ulcer lesions, stool occult blood ≥ (++), should not be included in the group; If fecal occult blood (+), gastroscopy is required；
9. Had an abdominal fistula, gastrointestinal perforation, or abdominal abscess in the 28 days prior to joining the study；
10. Patients with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds) who are prone to bleeding or are receiving thrombolytic or anticoagulant therapy；
11. Patients with central nervous system metastases or known brain metastases；
12. Patients with past and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function；
13. Urine routine showed urine protein ≥++ or confirmed 24 hours urine protein quantity > 1.0 g；
14. Severe thyroid disease cannot be controlled by treatment；
15. Rheumatic or autoimmune diseases, and immunosuppressant or high-dose hormone therapy after organ transplantation；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From Baseline to disease progress, up to 18 months
  Objective Response Rate was defined as the proportion of patients with a best objective response of complete response (CR) or partial response (PR) according to RECIST criteria (version 1.1).

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | From Baseline to primary completion date, about 2 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.
Progression free survival | From Baseline to primary completion date, about 2 years
  Progression-free survival is defined as the time from enrollment to the first documented disease progression according to RECIST version 1.1, or to death from any cause, whichever occurred first
Overal survival | From Baseline to primary completion date, about 5 years
  Time from randomization to death (from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Study Chair — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China